CLINICAL TRIAL: NCT07347366
Title: Effects of Electromagnetic High-Frequency Chest Wall Oscillation on Pulmonary Mucus Clearance in Patients With Impaired Self-Expectoration: An Investigator-Initiated, Single-Center, Prospective, Exploratory Study
Brief Title: Electromagnetic High-Frequency Chest Wall Oscillation on Pulmonary Mucus Clearance in Patients With Impaired Self-Expectoration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-2025-005
Record Dates: First submitted 2025-12-23; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Sputum
Keywords: sputum clearance; respiratory symptoms; Pulmonary Mucus Clearance; Electromagnetic High-Frequency Chest Wall Oscillation
MeSH Terms: conditions — Signs and Symptoms, Respiratory

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): A high-frequency chest wall oscillation device in the form of a vest (Todaki) is used in patients who require clearance of mucus retained in the lungs, providing high-frequency chest wall vibrations to dislodge sputum adherent to the bronchial walls and facilitate removal of secretions.
  Interventions: Device: CAREWAY
- Nine-Motor Device Group (Experimental): Description:This bed-type medical device delivers vibrational energy across the chest wall for patients with respiratory conditions. aiding in the clearance of accumulated sputum in the airways and lungs. It incorporates nine electromagnetic high-frequency, low-strain vibration motors to produce distributed vibrational energy, which is applied via the chest wall oscillation plate to multiple lung regions, enhancing comprehensive sputum clearance through multi-point oscillation
  Interventions: Device: EM HFLS CWSE(Nine-Motor)
- Single-Motor Device Intervention (Experimental): Description: This bed-type medical device applies vibrational energy to the chest wall of patients with respiratory diseases to facilitate sputum clearance from the airways and lungs. The device employs a single electromagnetic high-frequency, low-strain vibration motor that generates vibrational energy, which transmits through the chest wall oscillation plate directly to the patient's chest, promoting effective mucus mobilization via targeted oscillations.
  Interventions: Device: EM HFLS CWSE(Single-motor)

INTERVENTIONS:
Device: CAREWAY — CAREWAY , A high-frequency chest wall oscillation device in the form of a vest (Todaki) is used in patients who require clearance of mucus retained in the lungs, providing high-frequency chest wall vibrations to dislodge sputum adherent to the bronchial walls and facilitate removal of secretions.
  Arms: Control Group
Device: EM HFLS CWSE(Nine-Motor) — This bed-type medical device delivers vibrational energy across the chest wall for patients with respiratory conditions aiding in the clearance of accumulated sputum in the airways and lungs. It incorporates nine electromagnetic high-frequency, low-strain vibration motors to produce distributed vibrational energy, which is applied via the chest wall oscillation plate to multiple lung regions, enhancing comprehensive sputum clearance through multi-point oscillation
  Arms: Nine-Motor Device Group
Device: EM HFLS CWSE(Single-motor) — This bed-type medical device applies vibrational energy to the chest wall of patients with respiratory diseases , to facilitate sputum clearance from the airways and lungs. The device employs a single electromagnetic high-frequency, low-strain vibration motor that generates vibrational energy, which transmits through the chest wall oscillation plate directly to the patient's chest, promoting effective mucus mobilization via targeted oscillations.
  Arms: Single-Motor Device Intervention

SUMMARY:
This exploratory study aims to evaluate the efficacy and safety of an electromagnetic high-frequency, low-strain chest wall oscillation device for enhancing pulm

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients who require sputum clearance.
* Patients who present with fever or respiratory symptoms (cough, sputum) and, after confirmation of findings on imaging studies, are judged by the clinician to require sputum clearance.
* Adult patients (≥ 18 years) who have signed the informed consent form, or patients for whom consent has been obtained from a legally authorized representative

Exclusion Criteria:

* Patients with severe pneumonia requiring intensive care unit (ICU) treatment.
* Patients with major pulmonary diseases other than pneumonia, such as active tuberculosis or lung cancer.
* Patients with severe respiratory failure (PaO₂/FiO₂ ≤ 200 mmHg).
* Patients with hemodynamically unstable cardiovascular disease (myocardial infarction within the past 3 months, or heart failure of NYHA class 3 or higher).
* Patients hospitalized for head and neck trauma whose surgical site has not yet healed.
* Patients with serious cardiac arrhythmias or hemodynamic instability.
* Patients who have had pneumothorax or massive hemoptysis within the past 6 months, or who currently have hemoptysis.
* Patients who have undergone spinal surgery within the past 6 months or who have acute spinal injury.
* Patients with osteoporosis.
* Patients with bronchopleural fistula.
* Pregnant or breastfeeding women.
* Patients diagnosed with cervical disc disease.
* Individuals who have participated in clinical studies two or more times in the same year, or who have participated in another clinical study within the past 6 months (however, patients enrolled in chronic lung disease cohort studies such as asthma or COPD are allowed).
* Individuals who, in the judgment of the principal investigator or sub-investigator, have clinically significant findings that make them unsuitable for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
BCSS, Breathlessness, Cough, and Sputum Scale | Change rate in Breathlessness, Cough, and Sputum Scale (BCSS) scores at 1 week compared with baseline.
  The Breathlessness, Cough, and Sputum Scale (BCSS) is a patient-reported outcome measure assessing the severity of breathlessness, cough, and sputum. Each symptom is rated by the patient on a numeric scale from 0 (no symptoms) to 4 (severe symptoms). Individual symptom scores and the total score, calculated as the sum of the three items (range 0-12), are used for analysis, with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
mMRC (modified Medical Research Council Dyspnea Scale) | Change rate in modified Medical Research Council (mMRC) dyspnea scores at 1 week compared with baseline for patient symptom assessment.
  The modified Medical Research Council (mMRC) Dyspnea Scale is a patient-reported measure assessing the degree of breathlessness during daily activities. Dyspnea severity is rated on a 5-point ordinal scale ranging from 0 (breathlessness only with strenuous exercise) to 4 (too breathless to leave the house or breathless when dressing or undressing). Higher scores indicate more severe dyspnea.
St. George's Respiratory Questionnaire (SGRQ) | Change rate in St. George's Respiratory Questionnaire (SGRQ) scores at 1 week compared with baseline.
  The St. George's Respiratory Questionnaire (SGRQ) is a validated patient-reported outcome measure assessing health-related quality of life in patients with respiratory disease. It consists of three domains: Symptoms, Activity, and Impacts. Domain scores and the total score range from 0 to 100, with higher scores indicating worse health status and greater impairment of respiratory-related quality of life.
Visual Analog Scale for Dyspnea (VASD) | Scores at 1 week compared with baseline.
  It is a subjective assessment scale in which patients rate their perceived "difficulty in breathing" from 0 (none) to 10 (worst), and it is used to objectively assess changes in symptoms and evaluate treatment effects in patients with respiratory or cardiac diseases
VAS (Visual Analogue Scale) - Cough | Scores at 1 week compared with baseline.
  The severity of cough (VAS) is assessed using a Visual Analogue Scale, a subjective method in which patients rate the severity of their cough by marking their symptoms on a straight line from 0 (no cough at all) to 10 (the worst imaginable), which is then recorded as a score.
Cough And Sputum Assessment Questionnaire (CASA-Q) | Scores at 1 week compared with baseline.
  Cough and sputum were assessed using the Cough and Sputum Assessment Questionnaire (CASA-Q), which evaluates symptom severity and impact across four domains. Domain scores range from 0 to 100, with higher scores indicating less severe symptoms and lower disease impact.
Oxygen saturation (SpO2) | Data at 1 week compared with baseline.
  Oxygen saturation measured by pulse oximetry, defined as the percentage of hemoglobin saturated with oxygen in arterial blood. Values are expressed as a percentage (%), with higher values indicating better oxygenation status.
Forced Vital Capacity (FVC) | Data at 1 week compared with baseline.
  Forced vital capacity measured using pulmonary function testing, defined as the maximum volume of air forcibly exhaled after full inspiration. Values are recorded in liters (L).
Forced Expiratory Volume in 1 Second (FEV1) | Data at 1 week compared with baseline.
  Forced expiratory volume in one second measured using pulmonary function testing, defined as the volume of air forcibly exhaled in the first second of a forced expiration. Values are recorded in liters (L).
FEV1/FVC Ratio | Data at 1 week compared with baseline.
  The ratio of forced expiratory volume in one second to forced vital capacity measured using pulmonary function testing. Values are expressed as a percentage (%).
Forced Expiratory Flow 25-75% (FEF 25-75) | Data at 1 week compared with baseline.
  Forced expiratory flow between 25% and 75% of forced vital capacity measured using pulmonary function testing, reflecting airflow in the mid-portion of forced expiration. Values are recorded in liters per second (L/s).
Peak Expiratory Flow (PEF) | Data at 1 week compared with baseline.
  Peak expiratory flow measured using pulmonary function testing, defined as the maximum flow achieved during a forced expiration. Values are recorded in liters per minute (L/min).

CONTACTS AND LOCATIONS:
Locations (1):
- Rehab lab, Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea